CLINICAL TRIAL: NCT06391437
Title: Prevalence Of Vitamin A Deficiency In Critically Ill Children With Sepsis And Its Association With Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amany Mohammed El-Rebigi, MD, Lecturer of Pediatric and Neonatology, Benha University
Other Study IDs: RC17-4-2023
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Vitamin A Deficiency in Children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Sex- and age-matched approximate-health children without sepsis will be recruited as a control group.
  Interventions: Diagnostic Test: Extraction of blood sample
- Studied group: All pediatric Patients from 29 days to 16 years old who were admitted to the pediatric intensive care unit (PICU) with sepsis as defined by International pediatric sepsis consensus conference will be consecutively recruited in this study.
  Interventions: Diagnostic Test: Extraction of blood sample

INTERVENTIONS:
Diagnostic Test: Extraction of blood sample — Blood samples will be collected from all patients during the first 24 h of admission before enteral nutrition and/ or parenteral nutrition.

SUMMARY:
Aim of the work is to assess the prevalence of vitamin A deficiency in critically ill children with sepsis and the association between vitamin A deficiency and clinical outcomes

DETAILED DESCRIPTION:
Vitamin A plays an essential role in a large number of physiological functions that encompass vision, growth, reproduction, hematopoiesis, and immunity.

Despite major advances in the knowledge of vitamin A biology, its deficiency is still a serious public health problem that affects an estimated 127 million preschool children. In children, vitamin A deficiency results in increased risks of mortality and morbidity from infections, blindness and anemia. Many of these effects can be linked to the immunological functions of vitamin A.

Vitamin A modulates immunity through its active metabolite retinoic acid (RA), which acts on retinoid receptors in various cell types. Studies utilizing various animal models of vitamin A or retinoid receptor deficiency have revealed an integral role for RA in immunity and tolerance.

Retinoic acid (RA) has been reported to promote anti-inflammatory regulatory T cell (Treg) differentiation and inhibit interleukin (IL)-6-induced proinflammatory T helper 17 (Th17) cells, which could balance pro- and anti-inflammatory immunity.

Vitamin A deficiency (VAD ) is associated with adverse health outcomes due to an increased risk of infection in children. VAD could impact immunity at multiple levels, including disturbing the integrity of the gastrointestinal mucosal barrier, decreasing monocyte and natural killer (NK) cell numbers, and impairing the function of macrophages, dendritic cells, and neutrophils.

Sepsis, a life-threatening organ dysfunction caused by a dysregulated host response to infection, contributes to millions of deaths worldwide each year, with a mortality rate of more than 25%. Remarkably, sepsis is a common cause of death in children. The mortality of severe sepsis was reported to be as high as 34.6% in children.

As a public health problem, sepsis has posed a significant burden on extensive health care resources for many years. It is reported as a complicated immune disorder characterized by both a hyperinflammatory immune response in the early stage and immunosuppression in the later stage.

Most deaths from sepsis occur due to opportunistic pathogen superinfections or latent viral reactivation resulting from immunosuppression.

VA is an immunomodulatory, and its deficiency may cause an imbalance between pro- and anti-inflammatory factors and impaired immune function, which are found in sepsis. There is a biological rationale that VAD may be a contributing factor related to poor clinical outcomes in patients with sepsis. Importantly, VAD is highly prevalent in children, especially in preschool children. However, there is limited data regarding the correlation between VAD and sepsis, so we hypothesize that VAD may play an important role in the pathogenesis and progression of sepsis in children.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric Patients from 29 days to 16 years old who were admitted to the pediatric intensive care unit (PICU) with sepsis as defined by International pediatric sepsis consensus conference will be consecutively recruited in this study.

Sex- and age-matched approximate-health children without sepsis will be recruited as a control group.

Exclusion Criteria:

1. - Age > 16 years old.
2. - Premature infants and low birth weight infants.
3. - Children with underlying organ dysfunction, having received chemotherapy or radiotherapy, hematological malignancies, primary or acquired immunodeficiency.
4. - Children who discharged against medical advice with an uncertain prognosis.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This is a prospective study will be conducted from May 2023 to October 2023 in pediatric intensive care unit (PICU) at Benha university Hospital
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Severity of sepsis in pediatric patients with vitamin A deficiency | 1 month
  Severity of sepsis in pediatric patients with vitamin A deficiency
Clinical outcomes in septic pediatric patients with vitamin A deficiency | 1 month
  Length of hospital stay and mortality rate in pediatric patients with vitamin A deficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Cairo, Egypt